CLINICAL TRIAL: NCT01583348
Title: An Open Case Series About Technical Feasibility of Routine Intraoperative Cholangiography (IOC) During Elective Rigid-hybrid Transvaginal Natural Orifice Transluminal Endoscopic Cholecystectomy (tvNCC)
Brief Title: Technical Feasibility of Routine Intraoperative Cholangiography During Elective Rigid-hybrid Transvaginal Natural Orifice Transluminal Endoscopic Cholecystectomy
Status: Completed | Type: Observational
Sponsor: Cantonal Hosptal, Baselland (Other)
Responsible Party: Principal Investigator, Daniel Steinemann, MD, Principle Investigator, Cantonal Hosptal, Baselland
Other Study IDs: 45/12
Record Dates: First submitted 2012-04-20; First posted 2012-04-24 (Estimated); Last update posted 2013-04-30 (Estimated); Status verified 2013-04

CONDITIONS: Gallstone Disease
Keywords: transvaginal; NOTES; cholecystectomy; cholangiography; symptomatic gallstone disease
MeSH Terms: conditions — Cholelithiasis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Women with gallstones: 30 women with symptomatic gallstone disease with an indication for elective cholecystectomy
  Interventions: Procedure: Cholangiography during transvaginal rigid-hybdrid NOTES cholecystectomy

INTERVENTIONS:
Procedure: Cholangiography during transvaginal rigid-hybdrid NOTES cholecystectomy — During transvaginal rigid-hybrid NOTES cholecystectomy a intraoperative cholangiography is performed. After dissection of the Calot's triangle and distal clipping of the cystic duct, the cystic duct is incised and a regular cholangiography catheter is inserted. Contrast is injected and an image is obtained using an image-converter. After extraction of the catheter the cystic duct is clipped proximally. This intervention is performed in all patients included in the study.

SUMMARY:
While gold standard in the treatment of symptomatic gall stones is laparoscopic cholecystectomy with instruments introduced through multiple abdominal wall incisions, transvaginal access to the peritoneal cavity offers an alternative avoiding injury of the abdominal wall. Transvaginal hybrid-NOTES cholecystectomy has been demonstrated effective and safe. However it has not been demonstrated up-to-date if intraoperative cholangiography is feasible during such procedure. This observational case series describes success and technical feasibility of intraoperative cholangiography during transvaginal cholecystectomy. The investigators hypothesis is that cholangiography is feasible equal to conventional laparoscopic cholecystectomy.

ELIGIBILITY:
Inclusion Criteria:

* symptomatic gallstone disease
* age > 18 years
* written informed consent

Exclusion Criteria:

* age < 18 years
* not able to understand informed consent
* pregnancy
* vaginal atresia
* florid vaginal infection
* gynecological neoplasia
* allergy to Iod
* missing informed consents
* emergency procedure

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Women with symptomatic gallstone disease with an indication for elective cholecystectomy
Sampling Method: Non-Probability Sample
Enrollment: 33 (Actual)
Dates: Start 2012-04; Primary Completion 2012-10 (Actual); Study Completion 2013-04 (Actual)

PRIMARY OUTCOMES:
Number of patients with successful introduction of cholangiography catheter into cystic duct (yes/no) | intraoperative
  Was the introduction of the cholangiography catheter into the cystic duct successfull during transvaginal rigid-hybrid cholecystectomy.

SECONDARY OUTCOMES:
Time required for cholangiography | intraoperative
  From incision of the cystic duct to clipping of the cystic duct
Intraoperative complications | intraoperative
postoperative complications | within 6 weeks from surgery

CONTACTS AND LOCATIONS:
Overall Officials: Andreas Zerz, MD, Study Chair — Cantonal Hospital Baselland, Department of Surgery, Bruderholz, Switzerland; Daniel C Steinemann, MD, Principal Investigator — Cantonal Hospital Baselland, Department of Surgery, Bruderholz, Switzerland; Önder Ögredici, MD, Principal Investigator — Cantonal Hospital Baselland, Department of Surgery, Bruderholz, Switzerland
Locations (1):
- Cantonal Hospital Baselland, Bruderholz, Department of Surgery, Bruderholz, Basel-Landschaft, Switzerland